CLINICAL TRIAL: NCT02375724
Title: A RANDOMISED, DOUBLE BLIND, PLACEBO CONTROLLED, PARALLEL STUDY TO ASSESS THE BENEFITS OF ACLIDINIUM BROMIDE IN THE RELIEF OF COPD SYMPTOMS INCLUDING COUGH WHEN ADMINISTERED TO PATIENTS WITH COPD
Brief Title: BENEFITS OF ACLIDINIUM BROMIDE IN THE RELIEF OF COPD SYMPTOMS INCLUDING COUGH
Acronym: M-34273-46
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D6560C00001; 2014-004715-37 (EudraCT Number); M-34273-46 (Other: Clinical Trial Protocol Code)
Record Dates: First submitted 2015-02-26; First posted 2015-03-03 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — aclidinium bromide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aclidinium Bromide 400 μg (Experimental): Aclidinium Bromide 400 μg twice daily by inhalation
  Interventions: Drug: Aclidinium Bromide
- Placebo (Placebo Comparator): placebo twice daily by inhalation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aclidinium Bromide — Inhaled Aclidinium 400 μg twice per day by Eklira Genuair Inhaler
  Arms: Aclidinium Bromide 400 μg
Drug: Placebo — Inhaled dose-matched placebo, twice per day by Eklira Genuair Inhaler
  Arms: Placebo

SUMMARY:
The aim of the present study is to evaluate the effect of aclidinium bromide 400 μg BID compared with placebo on COPD symptoms in a symptomatic patients population with moderate COPD and chronic bronchitis, and particularly assess the effects in cough by using specific tools to assess the occurrence and impact of this relevant COPD symptom.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or non-pregnant, non-lactating female aged ≥40. Women of childbearing potential will follow specific study requirements.
2. Current or ex-cigarette smoker, with a smoking history of at least 10 pack-years
3. Patients with a clinical diagnosis of moderate COPD, with a post bronchodilator test available within 6 months prior to Visit 1 (Screening), with FEV1 ≥50% and <80% and FEV1/FVC <70%.
4. Symptomatic patients with a CAT≥10 at Screening and Randomisation Visit (Visit 1 and 2)
5. Clinical Diagnosis of Chronic Bronchitis (defined as "presence of cough and sputum production for at least 3 months in each of 2 consecutive years")
6. Patient who is eligible and able to participate in the trial and who consent to do so in writing after the purpose and nature of the investigation have been explained

Exclusion Criteria:

1. History or current diagnosis of asthma.
2. Patients who suffered from a moderate or severe COPD exacerbation in the last year prior to Visit 1 (Screening) or during the run-in period.
3. Patients who develop a respiratory tract infection within 6 weeks before Visit 1 (Screening) or during the run-in period.
4. Clinically significant respiratory and cardiovascular conditions thought to be contributing to cough or likely to interfere in the conduct of the study.
5. Patient who in the investigator's opinion may need to start a pulmonay rehabilitation program during the study and/or patients who started/finished it within 3 months prior to Screening Visit.
6. Use of long-term oxygen therapy.
7. Patients in non-stable treatment with angiotensin-converting enzyme inhibitors or opiates.
8. Patients in treatment with mucolytics, antihistamines, expectorants or antitussive drugs including over-the-counter medication.
9. Patient who does not maintain regular day/night, waking/sleeping cycles including night shift workers.
10. Patient with clinically relevant abnormalities in the results of the physical examination at Visit 1 (Screening)
11. Patient with a history of hypersensitivity reaction to inhaled anticholinergics,sympathomimetic amines, or inhaled medication or any component thereof (including report of paradoxical bronchospasm).
12. Patient with known narrow-angle glaucoma, symptomatic bladder neck obstruction, acute urinary retention, or patients with symptomatic non-stable prostatic hypertrophy.
13. Patient with known non-controlled history of infection with human immunodeficiency virus (HIV) and/or active hepatitis
14. Current diagnosis of cancer other than basal or squamous cell skin cancer
15. Patient with any other serious or uncontrolled physical or mental dysfunction
16. Patient with a history (within 2 years prior to Screening Visit) of drug and/or alcohol abuse that may prevent study compliance based on investigator judgment.
17. Patient unlikely to be cooperative or that can not comply with the study procedures
18. Patient treated with any investigational drug within 30 days (or 6 half-lives, whichever is longer) prior to Visit 1 (Screening).
19. Patient who intend to use any concomitant medication not permitted by this protocol or who have not undergone the required stabilization periods for prohibited medication.
20. Any other conditions that, in the investigator's opinion, might indicate the patient to be unsuitable for the study.

Ages: 40 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- Germany (6):
  - Research Site, Berlin
  - Research Site, Dortmund
  - Research Site, Frankfurt
  - Research Site, Frankfurt am Main
  - Research Site, Hanover
  - Research Site, Lübeck
- Hungary (6):
  - Research Site, Balassagyarmat
  - Research Site, Debrecen
  - Research Site, Komárom
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Százhalombatta
- Italy (2):
  - Research Site, Napoli
  - Research Site, Pisa
- Spain (7):
  - Research Site, Alicante
  - Research Site, Barcelona
  - Research Site, Hospitalet de Llobregat(Barcel
  - Research Site, Laredo
  - Research Site, Madrid
  - Research Site, Santiago(A Coruña)
  - Research Site, Seville
- United Kingdom (3):
  - Research Site, Manchester
  - Research Site, Northwood
  - Research Site, Sidcup

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized in 30 study sites in 5 countries Germany (10 sites), Hungary (6), Italy (2), Spain (9) and the United Kingdom (3)
  First patient was enrolled in March 2015 and last patient last visit was in November 2015
Pre-assignment Details: 300 patients were screened; 269 were assessed as eligible and were randomized into the study
  Thirty-one patients failed screening, with the main reason for screening failure being non-fulfilment of the inclusion or exclusion criteria (24 patients)
Groups:
- Aclidinium 400 μg: Aclidinium bromide 400 μg BID administered by Genuair® multidose dry powder inhaler
- Placebo: Placebo BID administered by Genuair® multidose dry powder inhaler
Period: Overall Study
Arm/Group | Aclidinium 400 μg | Placebo
Started | 135 | 134
Completed | 129 | 128
Not Completed | 6 | 6
Not completed — Lack of Efficacy | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aclidinium 400 μg | Placebo | Total
Number analyzed (Participants) | 135 | 134 | 269
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.0 (8.4) | 62.0 (9.1) | 62.0 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 50 | 107
  Male | 78 | 84 | 162

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Overall Exacerbations of Chronic Pulmonary Disease Tool-Respiratory Symptoms (E-RS) Total Score Over the 8 Week Study Period
Description: The EXACT-Respiratory Symptoms (E-RS) questionnaire was completed every evening The E-RS scale is an instrument comprising a subset of EXACT items to test the effect of treatment on the severity of respiratory symptoms in stable COPD Eleven of the 14-items of the EXACT questionnaire provides information about COPD symptoms: The E-RS Total Score is an aggregate of three domains: chest symptoms (derived sum of 3 items), cough and sputum (derived sum of 3 items) and RS-breathlessness (derived sum of 4 items); Individual scores were rated from 0 to 4 The E-RS Total score is based on a logit scoring system with conversion to a 0 (lowest score) to 100 scale (highest score) with higher scores indicating more severe symptoms
Time Frame: Baseline to Week 8
Population: Intent to treat (ITT) population defined as all randomized patients who took at least one dose of investigational medicinal product E-RS data were available for 131/135 patients receiving aclidinium and 133/134 receiving placebo
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | Aclidinium 400 μg | Placebo
Number analyzed (Participants) | 131 | 133
Score | -1.75 (0.342) | -0.73 (0.342)
Statistical Analysis 1: Comparison: Aclidinium 400 μg vs Placebo; Test type: Superiority or Other; p = 0.0306, Mixed Models Analysis; Baseline and age as covariates; treatment group, sex, visit, smoking-status and treatment group-by-visit interaction as fixed effect factors; Least squares mean difference = -1.02, 95% CI 2-sided [-1.94 to -0.10]

2. Secondary Outcome: Change From Baseline in Overall E-RS Cough and Sputum Domain Score Over the 8 Week Study Period
Description: The scale range of the 'cough and sputum' domain of the E-RS was 0-11, with higher scores indicating more severe symptoms
Time Frame: Baseline to Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | Aclidinium 400 μg | Placebo
Number analyzed (Participants) | 131 | 133
Score | -0.54 (0.090) | -0.33 (0.090)
Statistical Analysis 1: Comparison: Aclidinium 400 μg vs Placebo; Test type: Superiority or Other; p = 0.0793, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.22, 95% CI 2-sided [-0.46 to 0.03]

3. Secondary Outcome: Change From Baseline in the Leicester Cough Questionnaire (LCQ) Total Score at Week 8
Description: The LCQ is a self-administered questionnaire that assesses cough related quality of life The LCQ comprises 19 items and 3 domains (physical, psychological and social) The total score ranges from 3 to 21 and each domain scores range from 1 to 7; a higher score indicates a better quality of life
Time Frame: Week 8
Population: Intent to treat (ITT) population defined as all randomized patients who took at least one dose of investigational medicinal product LCQ data were available for 126/135 patients receiving aclidinium and 128/134 receiving placebo
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | Aclidinium 400 μg | Placebo
Number analyzed (Participants) | 126 | 128
Score | 1.18 (0.214) | 1.24 (0.214)
Statistical Analysis 1: Comparison: Aclidinium 400 μg vs Placebo; Test type: Superiority or Other; p = 0.844, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.06, 95% CI 2-sided [-0.64 to 0.52]

ADVERSE EVENTS:
Time Frame: Day 70±3
Arm/Group | Aclidinium 400 μg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/135 | 2/134
Other Adverse Events (participants affected / at risk) | 11/135 | 20/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aclidinium 400 μg (N=135) | Placebo (N=134)
Angina pectoris (Cardiac disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aclidinium 400 μg (N=135) | Placebo (N=134)
Headache (Nervous system disorders) | 7 | 13
Nasopharyngitis (Infections and infestations) | 4 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication and/or presentation whether complete or partial, of any part of the data or results of this trial will not be allowed until global publication and study results disclosure by the sponsor as per EMA / FDA regulatory compliance obligations, and only after mutual agreement between the investigator and the sponsor